CLINICAL TRIAL: NCT04238702
Title: A Randomized, Comparator-controlled, Cross-over Intervention Study to Assess Renal Hemodynamics of Mono- and Combination Therapy With SGLT-2 Inhibitor Empagliflozin and RAS-inhibitor Losartan in Patients With Type 2 Diabetes Mellitus
Brief Title: Renohemodynamic Effects of Combined empagliflOzin and LosARtan
Acronym: RECOLAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, D van Raalte, Principle Investigator, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DC2019RECOLAR01
Record Dates: First submitted 2019-09-11; First posted 2020-01-23 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Diabetes Mellitus, Type 2; Diabetic Kidney Disease
Keywords: RAS inhibition; Sodium Glucose Cotransport 2 inhibitors
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies | interventions — empagliflozin; Losartan

STUDY DESIGN:
Intervention Model Description: A phase 4, monocenter, randomized, double-blind, placebo-controlled, 4-armed cross-over mechanistic intervention study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Empagliflozin + Losartan (Experimental): Empagliflozin + Losartan
  Interventions: Drug: Empagliflozin 10 MG; Drug: Losartan 50Mg Tab
- Losartan + Placebo (Experimental): Losartan + Placebo
  Interventions: Drug: Losartan 50Mg Tab; Other: Placebo
- Empagliflozin + Placebo (Experimental): Losartan + Placebo
  Interventions: Drug: Empagliflozin 10 MG; Other: Placebo
- Placebo + Placebo (Placebo Comparator): Placebo + Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Empagliflozin 10 MG 7 days intervention period
  Other Names: Jardiance
  Arms: Empagliflozin + Losartan; Empagliflozin + Placebo
Drug: Losartan 50Mg Tab — Losartan 50 MG 7 days intervention period
  Other Names: Cozaar
  Arms: Empagliflozin + Losartan; Losartan + Placebo
Other: Placebo — Placebo 7 days intervention period
  Arms: Empagliflozin + Placebo; Losartan + Placebo; Placebo + Placebo

SUMMARY:
Worldwide, diabetic kidney disease (DKD) is the most common cause of chronic and end stage kidney disease. In parallel with the ever-increasing rates of obesity and type 2 diabetes (T2D), the incidence of DKD is expected to further increase in the coming years. DKD is a multi-factorial condition, involving pathophysiological factors such as chronic hyperglycemia, obesity, systemic- and glomerular hypertension, dyslipidemia, oxidative stress and pro-inflammatory cytokines. Large-sized prospective randomized clinical trials indicate that intensified glucose and blood pressure control, the latter especially by using agents that interfere with the renin-angiotensin-aldosterone system (RAS), halts the onset and (particularly) the progression of DKD, in both type 1 diabetes mellitus (T1DM) and T2DM patients. However, despite the wide use of angiotensin-converting enzyme (ACE) inhibitors and angiotensin receptor blockers (ARBs), a considerable amount of patients develop DKD, indicating an unmet need for renoprotective therapies. Sodium-glucose linked transporters (SGLT-2) inhibitors are a relatively novel glucose-lowering drug for the treatment of T2DM. These agents seem to exert pleiotropic actions 'beyond glucose control'. SGLT-2 inhibitors decrease proximal sodium reabsorption and decrease glomerular pressure and albuminuria in type 2 diabetes. In addition, SGLT-2 inhibitors reduce blood pressure and body weight. At this point in time, the renoprotective mechanisms involved with SGLT-2 inhibition still remain speculative, though a consistent finding is that SGLT-2 inhibitors reduce estimated eGFR after first dosing, which is reversible after treatment cessation. This "dip" indicates a renal hemodynamic phenomenon reminiscent of the RAS blockers and is thought to reflect a reduction in intraglomerular pressure. The potential renoprotective effects and mechanisms of combination therapy of SGLT-2 inhibitors and RAS inhibitors have not been sufficiently detailed in human type 2 diabetes. Therefore, the current study aims to explore the underlying mechanism of the improved renal hemodynamics and mechanistics of mono- and combination therapy with an SGLT-2 inhibitor and a RAS inhibitor on renal physiology in metformin and/or SU-treated T2DM patients.

DETAILED DESCRIPTION:
Diabetic kidney disease (DKD), characterized by reduced whole-kidney glomerular filtration rate (GFR) and/or urinary protein leakage, is a feared complication of type 2 diabetes (T2DM). With severe consequences such as endstage kidney disease (ESKD) and renal death, and strongly linked to cardiovascular (CV) morbidity and mortality, optimal treatment of DKD is vital. Still, even with multifactorial treatment of renal risk factors, including hyperglycemia, hypertension, obesity, dyslipidemia and albuminuria, residual risk remains high worldwide. Since the introduction of blockers of the renin-angiotensin-aldosterone system (RAS), no other renoprotective drug for T2D has been successfully developed, highlighting the need for novel strategies or new therapeutic drugs to improve renal outcome in T2DM.

In this regard, the introduction of the sodium glucose cotransporter (SGLT)2 inhibitors has been met with great enthusiasm. Designed to inhibit glucose reabsorption in the proximal tubule they induce glycosuria which indeed reduces hyperglycemia. More importantly, these drugs have shown remarkable benefits on CV disease and renal outcome in large CV safety trials in T2DM patients with high risk of or established atherosclerotic cardiovascular disease (CVD) as well as in patients with DKD. The first of these trials, the EMPAgliflozin cardiovascular outcome event trial in type 2 diabetes mellitus patients-Removing Excess Glucose (EMPA-REG OUTCOME), was reported in 2015 and demonstrated, next to risk reductions in CV outcomes, impressive reductions in the prespecified secondary renal outcome. In two subsequently reported CV safety trials conducted with canagliflozin (CANVAS-Program) and dapagliflozin (DECLARE-TIMI 58), these promising results indicating renal benefit were further strengthened. Recently, the results of a dedicated placebo-controlled trial with canagliflozin (CREDENCE) in DKD patients were reported. The study was terminated early due to overwhelming beneficial effects. Yet, at this point in time, the renoprotective mechanisms involved with SGLT2 inhibition still remain speculative, though a consistent finding is that SGLT2 inhibitors reduce estimated GFR after first dosing, which is reversible after treatment cessation. This "dip" indicates a renal hemodynamic phenomenon reminiscent of the RAS blockers and is thought to reflect a reduction in intraglomerular pressure. From studies in rodent models of type 1 diabetes (T1DM) and humans with type 1 diabetes it is hypothesized that SGLT2 inhibition leads to urinary sodium excretion by inhibiting in the proximal tubule, which influences renal hemodynamics through a mechanism known as tubuloglomerular feedback. In short, reduced sodium reabsorption at the level of the proximal tubule leads to increased sodium chloride delivery at the downstream located macula densa, which in turn increases afferent arteriolar resistance and reduces glomerular (hyper)filtration and hydrostatic pressure. In the recent RED trial (NCT02682563) the investigators assessed whether this is also true in T2DM patients. Suprisingly, this study showed that the renohemodynamic actions of SGLT2 inhibition in T2DM are not due to afferent vasoconstriction but rather efferent vasodilation. This is also the proposed working mechanism of inhibitors of the RAS system in T2DM, although dedicated studies in humans are scarcely done. Indeed, people with T2DM that do not respond to RAS blockers in terms of albuminuria reduction, also do not respond to SGLT2 inhibitor treatment.

Consequently, several questions remain regarding the combination of SGLT2 and RAS inhibitors. Especially with the recent results of CREDENCE, it is very likely that the combination of these agents will become standard of care in patients with T2DM and DKD. Both agents dilate the postglomerular arteriole, which might lead to relevant interactions or even synergistic effects. Since the majority of the population in the cardiovascular outcome trials used RAS inhibition, it is known that the renoprotective effect of SGLT2 inhibition is present with concurrent RAS inhibition. However, to what extend these agents interact and which of the various complex pathways involved in blood pressure and plasma volume control are affected by mono or combination therapy with these agents is unknown. It is important to emphasize that in the large trials, RAS blockade was not randomized and that the participants not on RAS blockade were small in numbers, making additional analyses on this topic difficult.

In conclusion: Despite multifactorial treatment approaches, residual risk for the development and progression of DKD remains high, and novel therapies or strategies to halt renal burden in T2DM are urgently needed. SGLT2 inhibitors and RAS inhibitors both induce glucose-independent renoprotective effects and improve renal outcome, seemingly via an at least partly equal mechanism, the dilation of the efferent glomerular arteriole resulting in an eGFR dip. The use of combination therapy with these agents could lead to an additive or even synergistic renoprotective effect in T2DM. As such, combined use of an SGLT2 inhibitor and RAS inhibitor may enhance individual benefits (e.g. reduction of glomerular pressure, activation of tubuloglomerular feedback, proximal and distal natriuresis, plasma volume contraction and reduction of blood pressure).

ELIGIBILITY:
Inclusion Criteria:

* Caucasian*
* Both genders (females must be post-menopausal; no menses >1 year; in case of doubt, Follicle-Stimulating Hormone (FSH) will be determined with cut-off defined as >31 U/L)
* Age: 35 - 80 years
* BMI: >25 kg/m2
* HbA1c: 6.5 - 10.0% Diabetes Control and Complications Trial (DCCT) or 48 - 86 mmol/mol International Federation of Clinical Chemistry (IFCC)
* Treatment with a stable dose of metformin and/or SU therapy for at least 3 months prior to inclusion
* Written informed consent

Exclusion criteria:

* History of unstable or rapidly progressing renal disease
* Macroalbuminuria; defined as ACR of 300mg/g.
* Estimated GFR <60 mL/min/1.73m2 (determined by the Modification of Diet in Renal Disease (CKD-EPI) study equation)
* Only use of alpha blockers is allowed as antihypertensive background therapy. Patients using an antihypertensive agent will be considered if this agent can be stopped (i.e. blood pressure adequate to stop at screening) or replaced by an alpha blocker. In these patients, a 4 week wash-out/run-in period will be observed prior to visit 2.
* Current/chronic use of the following medication: SGLT2 inhibitors, RAS inhibitors, TZD, GLP-1RA, DPP-4 inhibitors, glucocorticoids, immune suppressants, antimicrobial agents, chemotherapeutics, antipsychotics, tricyclic antidepressants (TCAs) and monoamine oxidase inhibitors (MAOIs). Subjects on diuretics will only be excluded when these drugs cannot be stopped for the duration of the study.
* Volume depleted patients. Patients at risk for volume depletion due to co-existing conditions or concomitant medications, such as loop diuretics should have careful monitoring of their volume status.
* Chronic use of non-steroidal anti-inflammatory drugs (NSAIDs) will not be allowed, unless used as incidental medication (1-2 tablets) for non-chronic indications (i.e. sports injury, head-ache or back ache). However, no such drug can be taken within a time-frame of 2 weeks prior to renal-testing
* History of diabetic ketoacidosis (DKA) requiring medical intervention (e.g. emergency room visit and/or hospitalization) within 1 month prior to the Screening visit.
* Current urinary tract infection and active nephritis
* Recent (<6 months) history of cardiovascular disease, including:

  * Acute coronary syndrome
  * Chronic heart failure (New York Heart Association grade II-IV)
  * Stroke or transient ischemic neurologic disorder
* Complaints compatible with neurogenic bladder and/or incomplete bladder emptying (as determined by ultrasonic bladder scan)
* Severe hepatic insufficiency and/or significant abnormal liver function defined as aspartate aminotransferase (AST) >3x upper limit of normal (ULN) and/or alanine aminotransferase (ALT) >3x ULN
* (Unstable) thyroid disease; defined as fT4 outside of laboratory reference values or change in treatment within 3 months prior to screening visit
* History of or actual malignancy (except basal cell carcinoma)
* History of or actual severe mental disease
* Substance abuse (alcohol: defined as >4 units/day)
* Allergy to any of the agents used in the study
* Individuals who are investigator site personnel, directly affiliated with the study, or are immediate (spouse, parent, child, or sibling, whether biological or legally adopted) family of investigator site personnel directly affiliated with the study
* Inability to understand the study protocol or give informed consent

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Glomerular Filtration Rate (GFR) | 7 days
  change in mGFR after 7 days of treatment using iohexol
Effective Renal Plasma Flow (ERPF) | 7 days
  change in ERPF after 7 days of treatment using iohexol

SECONDARY OUTCOMES:
Glomerular Hydrostatic Pressure | 7 days
  glomerular hydrostatic pressure which will be assessed by the Gomez formulae
Arteriolar resistance | 7 days
  arteriolar resistance which will be assessed by the Gomez formulae
Renal tubular function | 7 days
  Elektrolytes in urine
GFR trajectory | 7 days
  Creatinine clearance
Systemic hemodynamics | 7 days
  Bloodpressure
Autonomic nervous system activity | 7 days
  Heart rate variability
Vascular function | 7 days
  Arterial stiffness (Pulse Wave Analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel van Raalte, MD PhD, Principal Investigator — Amsterdam UMC, location VU Medical Center
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Natale P, Palmer SC, Navaneethan SD, Craig JC, Strippoli GF. Angiotensin-converting-enzyme inhibitors and angiotensin receptor blockers for preventing the progression of diabetic kidney disease. Cochrane Database Syst Rev. 2024 Apr 29;4(4):CD006257. doi: 10.1002/14651858.CD006257.pub2. PMID 38682786